CLINICAL TRIAL: NCT03284970
Title: Effect of Interferon Beta-1a SC 44 µg Three Times Weekly (Tiw) (Rebif) and Dimethyl Fumarate (DMF, Tecfidera) on Infections and Lymphocytes in Patients 50 Years or Older From a Single Center Chart Review
Brief Title: Retrospective Study to Determine Effect of Rebif and Tecfidera on Infections and Lymphocytes
Status: Completed | Type: Observational
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Other Study IDs: MS200136_0077
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Interferon beta-1a; Dimethyl fumarate; Rebif; Tecfidera; Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rebif (interferon beta 1a): This study will retrospectively collect the data from the subjects who had been treated with Rebif subcutaneously (SC) at a dose of 44 micro-grams three times a week.
- Tecfidera (dimethyl fumarate): This study will retrospectively collect the data from the subjects who had been treated with Tecfidera.

SUMMARY:
This study will be a single center, retrospective, pilot study to determine the effect of Rebif (interferon beta-1a) and Tecfidera (dimethyl fumarate) on infections on total lymphocyte counts, grade of lymphopenia, Cluster of Differentiation 4 (CD4) and Cluster of Differentiation 8 (CD8) counts and ratios in subjects aged 50 years and above with Relapsing-Remitting Multiple Sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

* RRMS subjects who have been treated with interferon beta 1a SC 44 micro-gram thrice a week and dimethyl fumarate in inpatient or outpatient settings during the period from January 1, 2015 to December 31, 2015.
* Subjects with at least one year of laboratory values post-index date to analyze lymphocyte counts, and CD4 and CD8 counts. The date of first blood draw for laboratory tests after January 1, 2015 will be defined as the subject's index date.

Exclusion Criteria:

- Subjects who have been on treatment for less than 1 year after their index date.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include subjects aged 50 years or older with relapsing RRMS, identified from a feasibility assessment conducted at a single center in United States, who were treated with either interferon beta-1a SC 44 micro-gram or dimethyl fumarate between January 1, 2015 to December 31, 2015.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects With One or More Infections | Up to 12 months

SECONDARY OUTCOMES:
Percentage of Subjects With One or More Serious Infections | Baseline, 6 Months, 12 Months
Percentage of Subjects With One or More Opportunistic Infections | Baseline, 6 Months, 12 Months
Number of Infections per Subject | Baseline, 6 Months, 12 Months
Number of Serious Infections per Subject | Baseline, 6 Months, 12 Months
Number of Opportunistic Infections per Subject | Baseline, 6 Months, 12 Months
Total Lymphocyte Levels | Baseline, 6 Months, 12 Months
Percentage of Subjects With Lymphopenia Grades I, II, III and IV | Baseline, 6 Months, 12 Months
Cluster of Differentiation 4 (CD4) and Cluster of Differentiation 8 (CD8) Counts | Baseline, 6 Months, 12 Months
Cluster of Differentiation 4 (CD4) and Cluster of Differentiation 8 (CD8) Ratio | Baseline, 6 Months, 12 Months
Occurrence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline, 6 Months, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (1):
- Neurology Center of New England, Foxborough, Massachusetts, United States